CLINICAL TRIAL: NCT06257056
Title: Closed Loop Neuromodulation for Treatment-refractory Schizophrenia: A Pilot Study
Brief Title: Deep Brain Stimulation for Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Lega (Other)
Responsible Party: Sponsor-Investigator, Bradley Lega, Associate Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0110
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Treatment-Refractory Schizophrenia
Keywords: Deep Brain Stimulation; Schizophrenia; Treatment Resistant Schizophrenia
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: Participants will undergo a maximum of two experimental sessions with ketamine and at least one with placebo. No participant will undergo more than two ketamine administration sessions.
  This is an overall 12-month feasibility and safety study. The first 8-months will be open-label bilateral DBS that targets a brain region within brain networks implicated in schizophrenia, which will be followed by a 4-month double-blind randomized discontinuation study. After 8 months, participants will enter a double blind (participant and rater) discontinuation study for 4-months to confirm the clinical benefit of DBS among responders. Final Go-No Go checkpoint occurs after final participants reaches the end of the 12-month study period. Participants will be randomized to either the ON or OFF stimulation phase for 2 months each. If randomization is initially in the ON phase, for the first 2 months, there will be no change in the stimulation settings.
Masking Description: The investigators propose a clinical trial involving 12-months open-label bilateral DBS in subjects with treatment refractory schizophrenia. The open label period is intended to ensure that maximal benefit can be achieved with the current proposed protocol.
  Following open label optimization, to control for possible placebo, each subject will enter a double blinded randomized discontinuation, intended to confirm clinical benefit of DBS among responders (4 months).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Randomized Discontinuation Period: OFF then ON DBS (Experimental): Subjects randomized to this arm are initially "OFF" DBS after the open label period then gradually decreased in their optimized setting's amplitude for 8 weeks and then "ON" DBS for 8 weeks.
  Interventions: Device: Abbott Laboratories Infinity™ implantable deep brain stimulation system
- Experimental: Randomized Discontinuation Period: ON then OFF DBS (Experimental): Subjects randomized to this arm are initially "ON" DBS with optimized stimulation settings for 8 weeks after the open label period and then "OFF" DBS with gradually decreasing amplitude for 8 weeks.
  Interventions: Device: Abbott Laboratories Infinity™ implantable deep brain stimulation system

INTERVENTIONS:
Device: Abbott Laboratories Infinity™ implantable deep brain stimulation system — Deep brain stimulation (DBS) refers to the process of delivering an electrical current to a precise location in the brain

SUMMARY:
There are three hypotheses proposed for this study: 1) Participants will report no unanticipated serious adverse events during the eight months of treatment. 2) Investigators will successfully model psychotic versus non-psychotic brain states using support vector machine (SVM) classifiers. 3) Participants specific brain stimulation parameters can induce a change in the brain state consistent with non-psychotic states as measured by classifier output. Hypotheses 1, 2, and 3 address safety and tolerability, efficacy, and the putative mechanism of successful treatment.

The overall objective is to use next generation Deep Brain Stimulation (DBS) combined with antecedent stereo electroencephalogram (SEEG) mapping to establish a new therapy for treatment-refractory schizophrenia given the limitations of current treatment modalities.

The primary objective is to demonstrate safety of acute and chronic network guided stimulation for treatment-refractory schizophrenia.

Exploratory Objectives:

1. Use intracranial mapping (SEEG) combined with pharmacological manipulation of psychotic states to create a protocol for participant specific deep brain stimulation to treat treatment-refractory schizophrenia.
2. Develop closed loop stimulation protocols to modify brain states during psychotic brain activity induced by low-dose ketamine administration.
3. Investigate the use of mnemonic similarity to characterize brain networks related to symptoms of treatment-refractory schizophrenia.
4. Treatment-related objectives: Record a reduction in psychotic symptoms, as well as an improvement in psychosocial function and cognition.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (non-pregnant) between ages 22 and 70;
2. Diagnostic and Statistical Manual of Mental Disorders (DSM) -5 diagnosis (assessed by Structured Clinical Interview for DSM-5 Axis I disorders SCID-5) of schizophrenia as the primary diagnosis.
3. Medically healthy, without any acute serious medical disorders
4. Treatment refractory and previous trials of treatment defined as: Demonstrated non-sustained response to at least two different antipsychotic drugs from two different chemical families. And demonstrated non-sustained response to at least either an electroconvulsive therapy (ECT) or a clozapine trial.
5. Suffering from active and ongoing psychotic symptoms of a continuous and aversive nature.
6. The PANSS must remain greater than or equal to 90 on two separate assessments (at initial screening and 1 week before surgery), over a 1-month period;
7. At least one item on the PANSS positive subscale is 5 or greater.
8. Normal brain MRI within 3 months of surgery;
9. Stable antipsychotic medication regimen for the month preceding surgery;
10. Normal thyroid stimulating hormone (TSH) level within 12 months of study entry;
11. Other medical conditions must be stable for at least 6 months;
12. Able and willing to give informed consent and agree to attend regular clinic visits for at least 12 months following surgery;
13. Able to have a treating psychiatrist or close relative present for discussions about the study and co-sign informed consent;
14. Willingness to sign Treatment Contract.
15. Participants with a family or caregiver support system to aid the participant throughout the study will be preferentially selected for inclusion.
16. For women of childbearing potential:

    1. Required to provide a negative pregnancy blood test during screening phase of the study, and during several additional timepoints throughout study participation.
    2. Obligated to use highly effective (those that when used alone or in combination, result in a low failure rate [i.e., less than 1 percent per year], when used consistently and correctly) methods of birth control throughout study participation.
    3. Will be allowed to participate in the study only after a confirmed menstrual period.
17. For men: Obligated to use highly effective (those that when used alone or in combination, result in a low failure rate [i.e., less than 1 percent per year], when used consistently and correctly) methods of birth control throughout study participation.

Exclusion Criteria:

1. Active alcohol or substance use disorder within 6 months, excluding nicotine; Urine drug test positive for illicit drugs;
2. Current substantial suicidal risk as defined by a plan or clear immediate intent for self-harm, or made a suicide attempt within the last year; or as identified as The Columbia Suicide Severity Rating Scale (C-SSRS),
3. Neurological/Medical condition that makes the participant, in the opinion of the surgeon, a poor surgical candidate (e.g., progressive neurodegenerative disorder, significant cardiopulmonary disorder, need for chronic anticoagulation);
4. Any history of seizure disorder, hemorrhagic stroke, or has high risk of seizure (history of congenital brain malformation, history of brain injury, neuro-developmental disorder, currently taking medication that is known to lower seizure threshold, or other factors that predispose seizures);
5. Any medical contraindication to surgery such as infection;
6. Coagulopathy: Bleeding propensity and/or one of the following: international normalised ratio (INR) > 1.5; prolonged activated partial thromboplastin time (aPTT) ≥ 45 sec; platelet count < 100×103 /uL;
7. Uncontrolled hypertension (systolic > 140mmHg and/or diastolic > 90 mmHg), demonstrated on each of three repeated measurements taken within one hour regardless of whether or not the participant is taking antihypertensive medications.
8. Patients with a heart-rate corrected QT interval (QTc) of > 450 msec
9. Participation in another drug, device, or biological study within 90 days;
10. Current implanted stimulation devices including cardiac pacemakers, defibrillators, and neurostimulators including spinal cord stimulators and deep brain stimulators;
11. Need for Diathermy;
12. Chronic use of anticoagulant or anti-platelet agents that cannot be safely stopped for a sufficient duration (minimum 2.5 weeks) in the peri-operative period.
13. Any Psychiatric/Neurological/Medical condition that makes the participant, in the opinion of the Investigator, a poor candidate.
14. A female participant of childbearing potential who is not able or willing to use highly effective (those that when used alone or in combination, result in a low failure rate [i.e., less than 1 percent per year], when used consistently and correctly) methods of birth control throughout the duration of participation in the trial.
15. A female participant of childbearing potential who is not able or willing to provide a negative pregnancy blood test during the screening phase of the study and during several additional timepoints throughout study participation. Specifically, the investigators will require a pregnancy test on the day of ketamine (or placebo) administration to avoid the risk of administering ketamine to a pregnant patient.
16. A separate cardiac condition that, in the opinion of study physician would present an unacceptable risk of undergoing general anesthesia or ketamine administration.
17. Participants with poorly controlled hypertension or persistent tachycardia, at baseline, will be excluded.
18. Participants who are taking an anti-depressant medication.
19. Any known contraindications for ketamine and/or esketamine (Spravato):

    1. Patients for whom a significant elevation of blood pressure would constitute a serious hazard, according to the opinion of the study PI.
    2. Patients with known hypersensitivity to ketamine, esketamine, or to any of the excipients.
    3. Patients with Aneurysmal vascular disease (including thoracic and abdominal aorta, intracranial, and peripheral arterial vessels) or arteriovenous malformation.
    4. Patients with a history of intracerebral hemorrhage.
    5. Patients with resting heart rate over 90 or below 55 beats per minute (BPM)
    6. Participants taking a medication with a known interaction with ketamine or esketamine (amphetamines, monoamine oxidase (MAO)-Is, aminophylline, theophylline, norepinephrine, epinephrine, vasopressin, dobutamine, ephedrine, ethanol, Ergometrine/Ergonovine). Patients taking benzodiazepines will not be excluded as this is recommended to prompt monitoring of patients in the information for esketamine. Dr. McDonagh will review such cases including for symptoms of sedation associated with their use and the dosage and duration of therapy for each. The investigators will exclude subjects who have any evidence of central nervous system (CNS) depression, such as decreased level of arousal or respiratory depression, thought to be linked with CNS depressants. The investigators will use the PRODIGY score to exclude any patient taking one of these medicines determined to be HIGH risk (score of 15 points or higher, https://www.apsf.org/wp-content/uploads/newsletters/online-only/202006/PRODIGY-Interactive-Risk-Assessment-Tool.pdf). The investigators note that ketamine has been used as an adjunct for sedation with benzodiazepines and opiates in the anesthesia environment, and the FDA's guidance on ketamine states: "KETALAR has been studied in over 12,000 operative and diagnostic procedures, involving over 10,000 patients from 105 separate studies. During the course of these studies KETALAR was administered as the sole agent, as induction for other general agents, or to supplement low-potency agents."
    7. During the ketamine administration phase in the hospital, patients with a history of benzodiazepine (or other CNS depressant) usage will undergo more frequent documentation of respiratory rate and heart rate (every 10 minutes). All patients will undergo continuous pulse oximetry monitoring to initiate supportive measures if there is any evidence of respiratory depression. In any patient with a history of opiate or 3-quinuclidinyl benzilate (BZ) administration, the investigators will have both flumazenil and naloxone immediately available at the bedside for administration if there is any evidence of respiratory distress.
    8. On the day of planned ketamine (or placebo) administration, Dr. McDonagh will review all medicines being administered to the patient to ensure there is no potential interaction. This will be documented on the Ketamine Administration Checklist included in appendix 6.
    9. On the day of planned ketamine (or placebo) administration, subjects will undergo a urine drug screen to avoid the accidental administration of ketamine to a patient who tests positive for any agents that is contraindicated (such as psychostimulants or CNS depressants). This is now reflected in the ketamine administration checklist (appendix 6).

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Demonstrate device safety | 3 years
  The primary objective is to demonstrate safety of acute and chronic network guided stimulation for treatment-refractory schizophrenia. This is determined if participants with the Deep Brain Stimulation Device demonstrate no significant device related serious adverse events (SAE).
  Device safety will be measured by number of reported SAE's in year 2 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Lega, M.D., Principal Investigator — University of Texas Southwestern Medical Center; David McDonagh, M.D., Principal Investigator — University of Texas Southwestern Medical Center; Nader Pouratian, M.D., Principal Investigator — University of Texas Southwestern Medical Center; Carol Tamminga, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Investigators with established research programs will be eligible for data sharing. Interested investigators will be required to submit a summary of proposed work and requested data elements. If approved by the Principal Investigator of the study, data will be shared. This data will be de-identified and coded. There is no plan to share identifiers outside the study team